CLINICAL TRIAL: NCT02888340
Title: A Randomized Controlled Trial of Acupuncture in the Emergency Department: A Pilot Study
Brief Title: Acupuncture in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S01022016
Record Dates: First submitted 2016-03-25; First posted 2016-09-05 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Pain
Keywords: Acupuncture; Emergency Department; Pain
MeSH Terms: conditions — Pain; Emergencies | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): One session of acupuncture prior to receiving pain medications after arriving to the emergency department with pain as a symptom.
  Interventions: Other: Acupuncture
- Usual Care (No Intervention): Usual care for pain, without intervention, after arriving to the emergency department with pain as a symptom.

INTERVENTIONS:
Other: Acupuncture — Acupuncture involves inserting thin, sterile needles into the skin. The needles do not go into the skin very far. Number of acupuncture sessions: one.
  Arms: Acupuncture

SUMMARY:
The investigators will study acupuncture in a pilot, randomized controlled trial (RCT) in the emergency department (ED) of a large, tertiary care hospital, Abbott Northwestern Hospital (ANW). The investigators suggest that the proposed intervention - provision of acupuncture in the ED as an alternative to usual ED care - will reduce pain and interrupt the trajectory (and potential cycle) of medication misuse by providing an alternative at a critical point of contact within the healthcare system, potentially disrupting the pathway from ED visit to opioid usage after discharge.

DETAILED DESCRIPTION:
The investigators will study acupuncture in a pilot, randomized controlled trial (RCT) in the emergency department (ED) of a large, tertiary care hospital, Abbott Northwestern Hospital (ANW). The investigators suggest that the proposed intervention - provision of acupuncture in the ED as an alternative to usual ED care - will reduce pain and interrupt the trajectory (and potential cycle) of medication misuse by providing an alternative at a critical point of contact within the healthcare system, potentially disrupting the pathway from ED visit to opioid usage after discharge. In this study, the investigators will assess the feasibility of implementation, practicality, and expansion of an acupuncture RCT in the ED environment. The study will prospectively measure and analyze change in pain intensity after treatment with acupuncture or usual care, use of opioids during ED visit, prescriptions written for opioids at ED discharge, and use of opioids at 30-day follow-up.

Study data will be collected using electronic health record (EHR) data and patient-reported outcomes. Patient-reported outcomes will be collected via an electronic database and solely for research purposes. The acupuncture intervention provided in the ED will be provided at no cost to the patient and will be paid for by the study sponsor. The practice of providing acupuncture in ANW's ED at no charge to the patient has been in place since November 2013. In conducting this pilot study, it will assess the ability to implement and carry out a RCT of acupuncture in the ED. By comparing pain change and opioid utilization among patients who receive acupuncture versus those who receive usual emergency department care, and by conducting follow-up data collection, the investigators will be able to better understand the potential role of a common non-pharmacological pain management strategy for mitigating pain and reducing opioid use in the emergency medicine setting.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Ability to communicate in English
* Non-critical status as determined at triage and / or by a clinic provider
* Presentation to the emergency department with acute musculoskeletal, back, pelvic, non-cardiac chest, abdominal, and headache pain (≥ 4 on the numerical rating scale), due to non-penetrating injury. Acute pain is defined by pain occurring within 72 hours of ED presentation (this can be an acute flare-up of a chronic pain condition).

Exclusion Criteria:

* Current pregnancy
* Need for emergent treatment as determined at triage and / or by a clinic provider (Level 1 or 2 on triage rating scale)
* Bone fracture
* Joint dislocation
* Fever exceeding 100° F
* Opioid medication taken orally within 4 hours (determined per patient report)
* Current use of a pharmaceutical analgesic patch
* Presenting with a chief complaint of a psychological / psychiatric concern
* Presenting with a migraine
* Having a unique treatment plan (UTP) on file with Abbott Northwestern Hospital
* Patient arriving via ambulance due to skipping triage
* Currently participating in this study due to previous ED admission
* Medical provider decision / clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-04; Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of delivering acupuncture via a Randomized Controlled Trial in the Emergency Department | At study completion, one year
  Assess feasibility of triaging and treating patients presenting to the emergency department with protocol defining criteria and then having that patient participate in a randomized controlled trial comparing acupuncture to usual care. This will be assessed by the number of patients approached compared to the number of patients consented and by the number of patients able to receive acupuncture while in the Emergency Department.

SECONDARY OUTCOMES:
Pain Reduction | During day 1 of study participation
  Measure pre- and post-treatment pain scores on an 11-point numerical rating scale for persons randomized to acupuncture or usual care in the emergency department. The goal of this outcome will be to obtain effect size to be used in the sample size calculation in a follow-up efficacy study.
Opioid use | At study completion, one year
  Collect information on opioid use in the emergency department, opioid prescriptions at discharge, and opioid medication usage at 30 days post-discharge in both the acupuncture and usual care arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reinstein AS, Erickson LO, Griffin KH, Rivard RL, Kapsner CE, Finch MD, Dusek JA. Acceptability, Adaptation, and Clinical Outcomes of Acupuncture Provided in the Emergency Department: A Retrospective Pilot Study. Pain Med. 2017 Jan 30;18(1):169-178. doi: 10.1093/pm/pnv114. PMID 26917627